CLINICAL TRIAL: NCT05026437
Title: The Value of CASUS vs. APACHE II in Predicting Mortality Among Patients Undergoing Coronary Artery Bypass Grafting
Brief Title: CASUS vs. APACHE II in Predicting Mortality After Coronary Artery Bypass Grafting
Acronym: CASUS
Status: Completed | Type: Observational
Sponsor: Antalya Training and Research Hospital (Other Government)
Collaborators: Dr. Siyami Ersek Thoracic and Cardiovascular Surgery Training and Research Hospital (Other); Haydarpasa Numune Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Sumeyye Ugur, drsumeyyeugur@gmail.com, Haydarpasa Numune Training and Research Hospital
Other Study IDs: SU2019
Record Dates: First submitted 2019-01-23; First posted 2021-08-30 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Coronary Artery Bypass Grafting; Mortality
Keywords: cardiac surgery score, mortality, ICU

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Cardiac surgery score and APACHE II scoring — Cardiac surgery score and APACHE II will calculated on the first postoperative day.

SUMMARY:
The study seeks to determine the value of CASUS in predicting mortality as compared with APACHE II scoring system among patients undergoing coronary artery bypass grafting.

DETAILED DESCRIPTION:
Patients undergoing coronary artery bypass grafting will prospectively studied after the admission to the cardiac intensive care unit. Data on the preoperative condition, intraoperative parameters, and postoperative course will collected. CASUS and APACHE II scores will calculated on the first postoperative day. Clinical outcomes are defined as 7-day mortality, 30-day mortality and morbidity. Morbidity includes variables such as length of stay in the cardiac surgical intensive care unit and in the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing coronary artery bypass grafting
* Over 18 years of age
* Staying at least 24 hours in the cardiac intensive care unit

Exclusion Criteria:

* Emergency surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population includes all adult patients who undergoing coronary artery bypass grafting during the study period.
Sampling Method: Probability Sample
Enrollment: 204 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2019-03-10 (Actual); Study Completion 2019-04-10 (Actual)

PRIMARY OUTCOMES:
Mortality at 7 days | 7 days
  Mortality in the first 7 days after surgery
Mortality at 30 days | 30 days
  Mortality in the first 30 days after surgery

SECONDARY OUTCOMES:
Length of stay in the cardiac intensive care unit | Up to 3 months (Through study completion)
  Only the length of the initial stay in the cardiac intensive care unit up to 3 months
Length of the stay in the hospital | Up to 3 months (Through study completion)
  It includes the period from surgery to discharge

CONTACTS AND LOCATIONS:
Overall Officials: Nihan YAPICI, Study Director — Dr. Siyami Ersek Thoracic and Cardiovascular Surgery TRH; Sümeyye UĞUR, Principal Investigator — Haydarpaşa Numune Training and Research Hospital
Locations (2):
- Turkey (Türkiye) (2):
  - Dr. Siyami Ersek Thoracic and Cardiovascular Surgery Training and Research Hospital in Turkey, Istanbul
  - Dr. Siyami Ersek Thoracic and Cardiovascular Surgery Training and Research Hospital, Istanbul

IPD SHARING:
Plan to Share IPD: Undecided